CLINICAL TRIAL: NCT05021159
Title: Assessing the Ontogeny of P-glycoprotein Expression in Blood of Pediatric Leukemic Patients
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Yasmine Elmorsi, Principal Investigator, Tanta University
Other Study IDs: 141052
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Acute Lymphocytic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Methotrexate Group: 20 acute lymphocytic leukemia patients receiving MTX treatment (3- 5 mg/ cm2)
  Interventions: Other: MTX, (but the investigator is not using any intervention, the participants are already taking it in their treatment protocol and the investigator is just analyzing p-gp expression)
- Healthy control group: 20 healthy pediatric subjects not receiving any treatment

INTERVENTIONS:
Other: MTX, (but the investigator is not using any intervention, the participants are already taking it in their treatment protocol and the investigator is just analyzing p-gp expression) — the investigator is not using any intervention, the participants are already taking it in their treatment protocol and the investigator is just analyzing p-gp expression
  Groups: Methotrexate Group

SUMMARY:
Determine P-glycoprotein expression in blood samples of Acute Lymphocytic leukemia (ALL) pediatric patients receiving MTX treatment and trace its ontogeny and compare it with its expression in pediatric healthy subjects. In addition, to determine the correlation of P-glycoprotein expression and Methotrexate concentration at steady state.

DETAILED DESCRIPTION:
The 20 leukemic patients will be classified into three age groups according to the ages that will be available at the time of sample collection.

* All patients will be recruited from Tanta Oncology Center, Tanta University.
* The study will be approved by the Research Ethics Committee of Tanta University and college of Pharmacy ethical committee.
* An informed consent will be obtained from parents of all patients in this research before enrollment.
* All patients' data will be private and confidential. Any unexpected risks that may appear during the course of the research will be reported to patients and the ethical committee on time.

Blood Samples will be obtained from healthy pediatric subjects of the same ages of the diseased group subjects (Samples will be obtained from subjects from a primary care center during their routine blood analysis excluding patients of chronic diseases, patients receiving any medications, and patients of impaired kidney or liver functions).

P-glycoprotein expression will be estimated in all samples using Permeability glycoprotein (P-gp), ELISA Kit, and its expression will be traced with development from the youngest till the oldest age available, this will also be compared with normal healthy pediatric subjects.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Acute Lymphocytic Leukemia Patients
* aged < 18 years old
* who are already taking the ALL MTX protocol.

Exclusion Criteria:

* Severe renal impairment (eGFR< 30 mL/min/1.73 m2 at screening)

  * Critically ill patients.
  * Other types of cancer

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric Acute Lymphocytic Leukemia Patients aged < 18 years old who are already taking the ALL MTX protocol.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
P-gp expression in blood samples | 42 hours
  P-gp expression in blood samples
Methotrexate concentration in blood samples | 42 hours
  Methotrexate concentration in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine M Elmorsi, Msc, Principal Investigator — Assistant lecturer in Clinical Pharmacy Dept., Faculty of pahrmacy, Tanta University; Osama M Ibrahim, Professor, Study Chair — Professor in Clinical Pharmacy Dept., Faculty of pahrmacy, Tanta University; Tarek M Mostafa, Professor, Study Chair — Assistant Professor in Clinical Pharmacy Dept., Faculty of pahrmacy, Tanta University
Locations (3):
- Egypt (3):
  - Faculty of Pharmacy, Tanta University, Tanta, Gharbia Governorate
  - Tanta Cancer Center, Tanta, Gharbia Governorate
  - Tanta University, Tanta, Gharbia Governorate

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aller SG, Yu J, Ward A, Weng Y, Chittaboina S, Zhuo R, Harrell PM, Trinh YT, Zhang Q, Urbatsch IL, Chang G. Structure of P-glycoprotein reveals a molecular basis for poly-specific drug binding. Science. 2009 Mar 27;323(5922):1718-22. doi: 10.1126/science.1168750. PMID 19325113
- [Background] Namanja HA, Emmert D, Davis DA, Campos C, Miller DS, Hrycyna CA, Chmielewski J. Toward eradicating HIV reservoirs in the brain: inhibiting P-glycoprotein at the blood-brain barrier with prodrug abacavir dimers. J Am Chem Soc. 2012 Feb 15;134(6):2976-80. doi: 10.1021/ja206867t. Epub 2011 Sep 9. PMID 21866921
- [Result] Kearns GL, Abdel-Rahman SM, Alander SW, Blowey DL, Leeder JS, Kauffman RE. Developmental pharmacology--drug disposition, action, and therapy in infants and children. N Engl J Med. 2003 Sep 18;349(12):1157-67. doi: 10.1056/NEJMra035092. No abstract available. PMID 13679531